CLINICAL TRIAL: NCT05859152
Title: Comparing the Outcomes of Intracytoplasmic Sperm Injection (ICSI) Using the Zona Pellucida-Bound Sperm Versus Conventional Manually Selected Sperm
Brief Title: Zona Pellucida Bound Sperm vs. Embryologist Selected Sperm for Intracytoplasmic Sperm Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IVIRMA-NorCal-Z01
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Infertility
Keywords: Intracytoplasmic Sperm Injection Procedure; ICSI
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP Bound Sperm Selection Oocyte Cohort (Experimental): This is half of the patient's mature oocytes that will be inseminated via the ICSI procedure with sperm that has bound to the ZP of an immature oocyte.
  Interventions: Other: Zona Pellucida-Bound Sperm Selection for ICSI
- Routine Care: Embryologist Selected Sperm Oocyte Cohort (Other): This is half of the patient's mature oocytes that will be inseminated via the ICSI procedure per routine with sperm that is subjectively selected by the embryologist (based on morphology and mobility characteristics). This is the current standard of care for ICSI.
  Interventions: Other: Routine Embryologist Selected Sperm

INTERVENTIONS:
Other: Zona Pellucida-Bound Sperm Selection for ICSI — one half of the patients' oocytes will be inseminated via the ICSI procedure with sperm that was bound to the ZP of an immature oocyte.
  Arms: ZP Bound Sperm Selection Oocyte Cohort
Other: Routine Embryologist Selected Sperm — one half of the patients' oocytes will be inseminated via the ICSI procedure with sperm that has been selected based on morphology and mobility characteristics by the embryologist per routine.
  Arms: Routine Care: Embryologist Selected Sperm Oocyte Cohort

SUMMARY:
This study aims to assess the clinical significance of the intracytoplasmic sperm injection (ICSI) with zona-pellucida (ZP) bound sperm compared to ICSI with embryologist selected sperm for patients undergoing in vitro fertilization treatment of their infertility.

DETAILED DESCRIPTION:
In this study, the investigators aim to determine the clinical utility of the ZP-bound sperm selection methodology for ICSI. This study will be a prospective, split cohort, randomized, control trial comparing the routine standard of sperm selection for ICSI via the embryologist versus sperm selected via ZP-binding for ICSI. Embryology, ploidy and clinical pregnancy outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing their first in vitro fertilization (IVF) cycle
* Electing single embryo transfer
* Electing preimplantation genetic testing for aneuploidy (PGT-A) of their embryos
* Female partners age <42 years old at start of vaginal oocyte retrieval cycle, but >18 years old.
* Normal ovarian reserve:
* Antimullerian hormone level (AMH) ≥ 1.2 ng/mL
* Antral follicle count (AFC) ≥ 8
* At least 4 mature oocytes (M2s) retrieved at the VOR procedure in order to randomize
* At least 1 immature oocyteretrieved at the VOR procedure to perform ZP binding co-incubation procedure
* Intention to transfer the morphological best quality, euploid, embryo at the frozen embryo transfer procedure

Exclusion Criteria:

* Contraindication to IVF
* Clinical indication for preimplantation genetic testing (i.e., screening for single gene disorder, chromosomal translocation, or any other disorders requiring a more detailed embryo genetic analysis)
* Male partner with azoospermia or oligozoospermia (<100,000 total motile spermatozoa)
* Male partner with Y-chromosome microdeletion
* Male partner with any Karyotype other than 46,XY
* Male partner requiring surgically obtained sperm either via testicular or epididymal retrieval procedures
* Uncorrected hydrosalpinges that communicate with the endometrial cavity
* Endometrial Insufficiency, as defined by a prior cycle with maximal endometrial thickness <6mm,), or persistent endometrial fluid
* Donor oocyte cycles
* Gestational carriers

Ages: 18 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Blastulation Rate | one week after the vaginal oocyte retrieval and ICSI procedure
  Blastulation rates per mature oocyte of ZP-bound versus embryologist selected sperm after ICSI.

SECONDARY OUTCOMES:
Fertilization Rate | 24 hours post ICSI procedure
  fertilization rates per mature oocyte of ZP-bound versus embryologist selected sperm after ICSI.
Blastocyst Ploidy Rate | Approximately 2 weeks after trophectoderm biopsy
  Preimplantation genetic testing for aneuploidy will be performed at the blastocyst stage and ploidy status compared between groups
Sustained Implantation Rates | Approximately 6 weeks after frozen embryo transfer procedure
  The number of participants discharged at 8-9 weeks gestational age to their obstetrician.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of Northern California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No